CLINICAL TRIAL: NCT00646425
Title: Randomized, Double-Masked, Placebo-controlled Evaluation of the Safety and Efficacy of Basiliximab as Maintenance Therapy in Subjects With Stable, Noninfectious Uveitis Who Undergo Tapering of Concomitant Immunosuppressive Medications
Brief Title: The Safety and Efficacy of Basiliximab as Maintenance Therapy in Subjects With Stable, Noninfectious Uveitis
Acronym: BSX-003
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cerimon Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Shaily Reichert, Cerimon Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSX-003
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Non-infectious Uveitis
Keywords: Non-infectious uveitis
MeSH Terms: interventions — Basiliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Basiliximab
  Interventions: Drug: Basiliximab
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Basiliximab — 40 mg basiliximab administered as short iv infusion once every 2 weeks for 3 doses and at Weeks 8 and 12 for a total of 5 doses
  Other Names: Simulect
  Arms: 1
Drug: Placebo — Placebo to match basiliximab
  Arms: 2

SUMMARY:
The objective of this trial is to assess if treatment with basiliximab allows subjects to taper off other immunosuppressive drug regimens without causing an increase in their uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of noninfectious intermediate, posterior or panuveitis of at least 3 months duration
* Treatment with greater than or equal to 20 mg/day of Prednisone at baseline or immunosuppressive drug score of greater than or equal to 5 at baseline
* BCVA by ETDRS protocol better than or equal to 20/200
* Intraocular pressure of 24 mmHg or less
* Anterior chamber cells and vitreous haze of less than or equal to 1
* Male or females, aged 12 or greater, body weight of 40 kg or greater

Exclusion Criteria:

* Prior treatment with Retisert
* Primary diagnosis of anterior uveitis, uveitis of infectious etiology or Behcet's disease
* Pregnancy or breast-feeding
* Increase in systemic immunosuppressive treatment regimen within 6 weeks before baseline

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To prevent an increase in disease activity as measured by anterior cell count, vitreal haze and visual acuity while subjects with stable noninfectious uveitis undergo tapering of concomitant immunosuppressive medications | The primary outcome will be assessed at Week 16

SECONDARY OUTCOMES:
Secondary objectives are to assess changes in visual acuity, retinal thickness, corticosteroid dose, and immunosuppressive drug score. Basiliximab pharmacokinetics and immunogenicity will also be assessed | These measures will be assessed at Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Shaily Reichert, Study Director — Cerimon Pharmaceuticals
Locations (6):
- United States (6):
  - Ocular Immunology & Uveitis Foundation, Cambridge, Massachusetts
  - Tauber Eye Center, Kansas City, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Southeast Clinical Research Associates, Belmont, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Vitreoretinal Consultants, Houston, Texas